CLINICAL TRIAL: NCT00580762
Title: Obesity, End-Stage Renal Disease and Kidney Transplantation
Brief Title: Bariatric Surgery for ESRD Patients vs Control
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Sanjay Kulkarni, Director of Kidney Transplantation, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0508000519
Record Dates: First submitted 2007-12-18; First posted 2007-12-27 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Obesity; ESRD
MeSH Terms: conditions — Obesity; Kidney Failure, Chronic | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ESRD (Experimental): End-Stage Renal Disease (ESRD) patients on dialysis who meet the NIH guidelines and preoperative requirements for RYGB will undergo laparoscopic RYGB
  Interventions: Procedure: Roux-en-y gastric bypass (RYGB)
- Non-ESRD (Active Comparator): Non-ESRD patients who meet the NIH guidelines and preoperative requirements for RYGB will undergo laparoscopic RYGB
  Interventions: Procedure: Roux-en-y gastric bypass (RYGB)

INTERVENTIONS:
Procedure: Roux-en-y gastric bypass (RYGB)

SUMMARY:
This study will address a true clinical problem by developing a risk/benefit analysis for rapid surgical weight loss in the ESRD population. The risks of surgical intervention, as well as, potential nutritional concerns, balanced with that of the potential medical benefits associated with significant weight loss.

DETAILED DESCRIPTION:
The study will be designed to compare two cohorts of patients that will undergo laparoscopic RYGB. Cohort 1 will include ESRD patients on HD who meet the NIH guidelines and preoperative requirements for RYGB. Cohort 2 will include non-ESRD patients who meet the NIH guidelines and preoperative requirements for RYGB. Laparoscopic RYGB will be performed in ESRD patients who meet the guidelines recommended by the National Institutes of Health consensus statement . This includes patients who either have a BMI≥40 kg/m2 or have a BMI≥35 kg/m2 and have a significant morbidity attributed to their obesity (i.e. sleep apnea, hypertension, and diabetes mellitus). All patients will undergo a complete pre-operative evaluation inclusive of dietary instruction, assessment of surgical risk, psychosocial evaluation and compliance evaluation. This evaluation will be conducted through an existing infrastructure at the investigators Bariatric Surgery Center. Patients will be required to be on hemodialysis or able to be converted to hemodialysis for the perioperative period. All procedures will be performed by the same team of surgeons, experienced in both laparoscopic RYGB, organ transplantation and general surgery in ESRD patients. The risks involved with Roux-en-Y gastric bypass surgery will be discussed with the patient. These risks are inherent to the procedure, however the procedure is being conducted for medical appropriate reasons and therefore the benefits to the procedure outweigh the risks. At the present time, it is believed, without any justification, that this procedure is more risky or too risky in the ESRD population. A primary objective of this study is to investigate this question.

ELIGIBILITY:
Inclusion Criteria:

1. Obese ESRD patients with a BMI≥ 40kg/m2 or ≥35kg/m2 with an medical complication attributed to morbid obesity (NIH guidelines).REF
2. Age ≥ 18 and ≤ 65
3. Patients must be on hemodialysis for one month.
4. Patients listed for kidney transplant in a UNOS certified kidney transplant center.
5. Patients have accrued less than 18 months of waiting time.
6. Completion of pre-RYGB psychosocial evaluation.
7. Completion of pre-RYGB dietary counseling.
8. Completion of pre-RYGB surgical risk assessment inclusive of cardiac evaluation.
9. Full reciprocal understanding of informed consent and the risks and benefits of RYGB procedure.
10. Acceptance of clinical protocol evaluations requiring scheduled clinic visits and laboratory blood draws.

Exclusion Criteria:

1. Age < 18 and > 65.
2. Patients with a history of peritoneal dialysis related bacterial peritonitis.
3. Peritoneal dialysis patients not willing to undergoing temporary hemodialysis.
4. History of difficult vascular access as defined by the inability to obtain permanent upper extremity or temporary jugular venous access.
5. History of poor hemodialysis performance.
6. Patients enrolled in another study within 6 months of initiation.
7. Patients listed for kidney transplant in a different UNOS region that has shorter transplant waiting times than the region governing the investigators institution.
8. Patients unwilling to be made temporarily unavailable for transplant.
9. History of non-compliance with medical care.
10. Uncontrolled psychiatric illness (ie. depression, anxiety, attention deficit disorder (ADD), uncontrolled binge eating disorder)
11. Inability to provide reciprocal understanding of informed consent.
12. Failure to complete the preoperative work-up (psychosocial, dietary and surgical risk) for RYGB.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The safety and efficacy of laparoscopic RYGB in obese ESRD patients will be assessed. | 1 year

SECONDARY OUTCOMES:
Weight reduction in ESRD patients will be characterized to assess additive risk factors for micronutrient abnormalities and protein malnutrition. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kulkarni, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States